CLINICAL TRIAL: NCT02469350
Title: Feasibility and Acceptability Study of Serious Game Rehabilitation Program in Parkinson's Disease Patients With Resistant Gait and Balance Disorders
Brief Title: Serious Game for Parkinson's Disease Patients
Acronym: PARKGAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C15-12; RCB (Registry Identifier: 2015-A00277-42)
Record Dates: First submitted 2015-05-28; First posted 2015-06-11 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease
Keywords: Gait and balance disorders; serious game
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation with serious game (Experimental): 18 rehabilitation sessions with serious game during a 6-8 weeks period
  Interventions: Other: Serious game

INTERVENTIONS:
Other: Serious game — Rehabilitation with serious game

SUMMARY:
In this study the investigators aim to assess the feasibility and acceptability of a serious game to rehabilitate gait and balance disorders in 10 patients with Parkinson's disease previously operated for deep brain stimulation of the sub thalamic nucleus.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Gait and balance disorders
* Chronic bilateral deep brain stimulation of the subthalamic nucleus (> 1 year).

Exclusion Criteria:

* Dementia
* Ongoing severe medical condition that prevented assessments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Feasibility questionnaire | once a week
  self-assessment questionnaire

SECONDARY OUTCOMES:
Acceptability questionnaire | once a week
  self-assessment questionnaire
biomechanical parameters of gait and balance | at inclusion, 3 weeks, 6 weeks and 18 weeks
  recordings of centres of foot and mass displacements and velocities
kinematics parameters of gait and balance | at inclusion, 3 weeks, 6 weeks and 18 weeks
  range of motion of hip, knee and ankle angles

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure Welter, MD, PhD, Principal Investigator — GHPS, APHP, Paris
Locations (1):
- ICM, CIC Neurosciences, Paris, France

REFERENCES:
- [Result] Nuic D, Vinti M, Karachi C, Foulon P, Van Hamme A, Welter ML. The feasibility and positive effects of a customised videogame rehabilitation programme for freezing of gait and falls in Parkinson's disease patients: a pilot study. J Neuroeng Rehabil. 2018 Apr 10;15(1):31. doi: 10.1186/s12984-018-0375-x. PMID 29636105